CLINICAL TRIAL: NCT00938795
Title: Uncertainty Management Intervention for Patients Awaiting Liver Transplant
Brief Title: Uncertainty Management Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00007468; 1P01NR010948-01 (NIH)
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Liver Diseases
Keywords: liver disease; uncertainty; self management
MeSH Terms: conditions — Liver Diseases | interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Uncertainty Management Intervention (Other): The Uncertainty Management Intervention will consist of six 30-minute phone calls with a study educator to discuss issues of psychological distress, uncertainty management, symptom control, self efficacy for symptom management, and quality of life.
  Interventions: Other: Uncertainty Management Intervention
- Comparison Conditions for Liver Disease (Other): Six 30-minute telephone calls that provide structured education about liver disease.
  Interventions: Other: Comparison Conditions for Liver Transplant

INTERVENTIONS:
Other: Uncertainty Management Intervention — Six 30-minute telephone calls with a nurse to discuss emotional and physical aspects of liver disease and awaiting liver transplant
  Arms: Uncertainty Management Intervention
Other: Comparison Conditions for Liver Transplant — Six 30-minute telephone calls that provide structured education about liver disease.
  Arms: Comparison Conditions for Liver Disease

SUMMARY:
The goal of this study is to improve symptoms and quality of life for end-stage liver disease patients awaiting a liver transplant and their caregivers by providing them with the resources and tools to self-manage their complex concerns.

DETAILED DESCRIPTION:
Hepatitis C Virus is the most common blood-borne infection in the U.S., affecting at least 4 million individuals, with more than 19,000 new cases occurring each year. Further, the CDC has projected a fourfold increase in the number of chronic hepatitis C patients between 1990 and 2015, and these patients are at risk for developing end stage liver disease (ESLD). By 2015 an estimated 375,000 chronic hepatitis C patients will develop cirrhosis and progress to ESLD, representing the majority of individuals who need liver transplants. ESLD is a life-limiting illness, and patients are told that, without a liver transplant, they may die.

This 5 year randomized controlled trial will test the efficacy of an Uncertainty Management Intervention delivered via telephone by a nurse to the patient and caregiver. An attention control group of patients and caregivers will receive phone calls to discuss their experience of awaiting a liver transplant. Based on the problems and concerns of patients waiting for a liver transplant and the prior success of the Intervention for patients dealing with serious chronic illness, we believe the Uncertainty Management Intervention adapted specifically for ESLD patients will lead to significant improvements in patients' and caregivers' abilities to manage the symptoms and distress associated with ESLD and the process of awaiting liver transplant.

The specific aims are to: 1) examine the effects of the Uncertainty Management Intervention on patient outcomes of psychological distress, uncertainty management, symptom control, self efficacy for symptom management, and QOL compared to an attention control group receiving calls to discuss their disease experience; 2) explore the effects of the Intervention on caregiver outcomes of uncertainty management, self-efficacy for helping the patient manage symptoms, and better QOL compared to an attention control group; 3) identify characteristics of individuals for whom the intervention is particularly effective.

Waiting for a liver transplant under conditions of uncertainty is a harrowing experience for patients and caregivers, yet there have been few attempts to test nursing interventions for ESLD patients. The overall goal of this project is to provide these patients and their caregivers the tools to self-manage their complex concerns. The anticipated outcome is ESLD patients awaiting liver transplant benefit from the Uncertainty Management Intervention, thus providing new knowledge for practitioners and policy makers.

ELIGIBILITY:
Inclusion Criteria (patient):

* Diagnosis of ESLD and on the liver transplant waiting list
* Receiving care at a Liver Clinic in the United States
* 18 years of age or older
* MELD greater than or equal to 11
* Able to read and speak English
* No major cognitive impairment
* Not a recipient of a prior transplant (any organ)
* Has a caregiver willing to participate

Inclusion Criteria (caregiver):

* 18 years of age or older
* Able to read and speak English
* Provides care to a patient meeting the above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2010-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Uncertainty Management | Five months

SECONDARY OUTCOMES:
Symptom control | Five months
Quality of life | Five months
Psychological distress | Five months

CONTACTS AND LOCATIONS:
Overall Officials: James Tulsky, MD, Principal Investigator — Duke University School of Nursing; Donald Bailey, PhD, Principal Investigator — Duke University School of Nursing; Annette Devito Dabbs, PhD, RN, Principal Investigator — The University of Pittsburgh; Paul H. Hayashi, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Laurel Williams-Salonen, RN,MSN,CCTC, Principal Investigator — The University of Nebraska Medical Center
Locations (4):
- United States (4):
  - The University of Nebraska Medical Center, Omaha, Nebraska
  - University of North Carolina-Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - The University of Pittsburgh, Pittsburgh, Pennsylvania